CLINICAL TRIAL: NCT00171665
Title: Efficacy and Safety of Diclofenac Sodium Gel in Hand Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VOSG-PE-315
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Osteoarthritis
Keywords: Hand osteoarthritis, Topical NSAID, Diclofenac sodium
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Drug: Diclofenac topical sodium gel 1%

SUMMARY:
This study will test the efficacy and safety of topical diclofenac sodium gel in the treatment of hand osteoarthritis.

ELIGIBILITY:
Key Inclusion criteria:

• Osteoarthritis of the hand

Key Exclusion Criteria:

* Other rheumatic disease, such as rheumatoid arthritis
* Active gastrointestinal ulcer during the last year
* Known allergy to analgesic drugs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2005-05; Study Completion 2005-12

PRIMARY OUTCOMES:
OA pain intensity in target hand at Week 4 and 6
Total AUSCAN score in target hand at Week 4 and 6
Global rating of disease activity by patient at Week 4 and 6

SECONDARY OUTCOMES:
OA pain intensity and total AUSCAN score in target hand, and global rating of disease activity by patient at Weeks 1, 2 and 8
AUSCAN pain, stiffness and physical function scores in target hand, and global rating of benefit by patient at Weeks 1, 2, 4, 6 and 8
OA pain intensity in target hand and use of rescue medication recorded in diary
Global evaluation of treatment at final visit
Treatment responder rate according to OARSI criteria

CONTACTS AND LOCATIONS:
Locations (69):
- United States (69):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - MedSearch, LLC, Calera, Alabama
  - Montgomery Rheumatology Associates, Montgomery, Alabama
  - Drug Research & Analysis Corp, Montgomery, Alabama
  - Arizona Center for Clinical Research, Glendale, Arizona
  - Quality of Life Medical Research Center, LLC, Tucson, Arizona
  - Lovelace Scientific Resources, Inc., Beverly Hills, California
  - Med Investigations/Med Center, Carmichael, California
  - H. Richard Barthel,MD, Inc., Santa Barbara, California
  - Clinical Research of CT/NY, Danbury, Connecticut
  - Allergy and Arthritis Associates, Hamden, Connecticut
  - Arthritis & Osteoporosis Center, PC, Hamden, Connecticut
  - Clinical Research Consultants, Stratford, Connecticut
  - Health Core, Newark, Delaware
  - Clinical Research of West Florida, Clearwater, Florida
  - The Community Research of South Florida, Hialeah, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Miami Research Associates, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Arthritis Research of Florida, Inc., Palm Harbor, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Andres Patron, DO PA, Pembroke Pines, Florida
  - Coastal Medical Research, Port Orange, Florida
  - University Neurology, Sarasota, Florida
  - Southwest Florida Clinical Research Center, Tampa, Florida
  - Radiant Research - Atlanta West, Atlanta, Georgia
  - Intermountain Orthopaedics, Boise, Idaho
  - Allan B. Aven, MD, SC, Arlington Heights, Illinois
  - Heartland Research Associates, LLC, Arkansas City, Kansas
  - Chesapeake Medical Research, LLC, Baltimore, Maryland
  - Arthritis Associates, Inc., Peabody, Massachusetts
  - Clinsite, Ann Arbor, Michigan
  - Twin Cities Clinical Research, Brooklyn Center, Minnesota
  - Radiant Research - Minneapolis, Edina, Minnesota
  - PrimeCare Research Associates, Florissant, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Comprehensive Clinical Research, Turnersville, New Jersey
  - Unifour Medical Research Associates, Hickory, North Carolina
  - Crescent Medical Research, Salisbury, North Carolina
  - Carolina Clinical Research, Winston-Salem, North Carolina
  - Wells Institute for Heatlh Awareness, Kettering, Ohio
  - Clinical Research Source, Perrysburg, Ohio
  - PRO Research, Eugene, Oregon
  - Allegheny Pain Management, Altoona, Pennsylvania
  - Neshaminy Medical, PC, Bensalem, Pennsylvania
  - Medical Group @ Marple Commons, Broomall, Pennsylvania
  - Westminster Family Medicine, Erie, Pennsylvania
  - Feasterville Family Health Care Center, Feasterville, Pennsylvania
  - Southeastern Pennsylvania Medical Institute, Havertown, Pennsylvania
  - Radiant Research, Philadelphia, Pennsylvania
  - Radiant Research - Reading, Wyomissing, Pennsylvania
  - Partners in Clinical Research, Woonsocket, Rhode Island
  - Radiant Research - Anderson, Anderson, South Carolina
  - Palmetto Medical Research, Mt. Pleasant, South Carolina
  - Harmony Research, Inc., Johnson City, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Amarillo Center for Clinical Research, Amarillo, Texas
  - Walter F. Chase, MD, PA, Austin, Texas
  - Quality Research, Inc., San Antonio, Texas
  - Radiant Research - San Antonio Northeast, San Antonio, Texas
  - Radiant Research - San Antonio, San Antonio, Texas
  - Texas Research Center, LLP, Sugar Land, Texas
  - Intermoutain Clinical Research, Salt Lake City, Utah
  - Radiant Research - Salt Lake City, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Radiant Research - Tacoma, Lakewood, Washington
  - Advanced Healthcare, SC, Milwaukee, Wisconsin
  - Dean Medical Center - Oregon Clinic, Oregon, Wisconsin

REFERENCES:
- [Derived] Barthel HR, Peniston JH, Clark MB, Gold MS, Altman RD. Correlation of pain relief with physical function in hand osteoarthritis: randomized controlled trial post hoc analysis. Arthritis Res Ther. 2010;12(1):R7. doi: 10.1186/ar2906. Epub 2010 Jan 11. PMID 20064249
- [Derived] Altman RD, Dreiser RL, Fisher CL, Chase WF, Dreher DS, Zacher J. Diclofenac sodium gel in patients with primary hand osteoarthritis: a randomized, double-blind, placebo-controlled trial. J Rheumatol. 2009 Sep;36(9):1991-9. doi: 10.3899/jrheum.081316. Epub 2009 Jul 31. PMID 19648310